CLINICAL TRIAL: NCT03858153
Title: The Effects of Exercise and Nutrition Interventions on Chemotherapy-induced Peripheral Neuropathy and Interoceptive Brain Circuitry
Brief Title: Exercise and Nutrition Interventions During Chemotherapy K07
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Po-Ju Lin, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00003387; K07CA221931 (NIH)
Record Dates: First submitted 2019-02-15; First posted 2019-02-28 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neuropathy;Peripheral
Keywords: chemotherapy
MeSH Terms: conditions — Neuritis | interventions — Nutrition Assessment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor and investigator will be masked of Arms to the extent possible (i.e., for some outcomes e.g., biomarkers but not others e.g. symptom tests).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Exercise for Cancer Patients (EXCAP©®) involves face-to-face instruction and a prescription for an at-home progressive walking and resistance exercise program.
  Interventions: Behavioral: EXCAP Exercise
- Nutrition Education (Active Comparator): Nutrition education involves equal time and attention as the exercise arm, but the content covers nutrition for cancer patients and lacks an exercise prescription.
  Interventions: Behavioral: Nutrition Education

INTERVENTIONS:
Behavioral: EXCAP Exercise — 12 weeks of at-home walking and resistance exercise.
  Arms: Exercise
Behavioral: Nutrition Education — 12 weeks of implementing eating tips and tracking food.
  Arms: Nutrition Education

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN) is a highly prevalent and severe side-effect of taxane chemotherapy, often used to treat breast cancer. Unfortunately there are very limited treatments for CIPN. This is a phase II randomized controlled trial to test the preliminary efficacy of exercise vs. nutrition education on CIPN, to systematically investigate the potential roles of inflammation and interoception, and to obtain data with a more accurate effect size to inform a future study.

ELIGIBILITY:
Inclusion criteria (subjects must…)

1. Be female
2. Have breast cancer
3. Be scheduled to receive taxane chemotherapy without other neurotoxic chemotherapy (platinums, vinca alkaloids, bortezomib, thalidomide)
4. Have at least six months life expectancy according to the patient's oncologist or designee
5. Be able to read English
6. Be at least 18 years old (no upper limit on age)
7. Provide written informed consent

Exclusion criteria (subjects must not…)

1. Be in the active or maintenance stage of exercise behavior (i.e., subjects must be sedentary)
2. Have physical limitations (e.g., cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in maximal physiological fitness testing and a low/moderate intensity home-based walking and progressive resistance exercise program.

Additional exclusion criteria only for patients performing the MRI scanning (40 of 80 enrolled subjects)

1. Subjects must not have contraindications for MRI scanning (pacemaker, metal implants, pregnancy, chest expander from breast reconstruction, etc.-note that most port-a-caths are safe for MRI scanning)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-08-27 (Actual)

PRIMARY OUTCOMES:
Patient-reported sensory symptoms of chemotherapy-induced peripheral neuropathy (CIPN) | Time point 2 (approximately 6 weeks), controlling for baseline value
  CIPN-20 sensory subscale (Postma et al 2005). The subscale includes 9 questions, each rated 1-4, and the score ranges from 9-36 with larger values reflecting more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).

SECONDARY OUTCOMES:
Sensory loss | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Finger tactile sensitivity
Numbness and tingling | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Patient-reported severity of numbness/tingling (0-10). A larger value reflects more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).
Sensory, motor, and autonomic symptoms of CIPN | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks) or time point 4 (approx. 24 weeks), controlling for baseline
  CIPN-20 total score (Postma et al 2005). The score includes 20 questions, each rated 1-4, and the score ranges from 20-80 with larger values reflecting more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).
Patient-reported sensory symptoms of CIPN | Time point 3 (approx. 12 weeks) or time point 4 (approx. 25 weeks), controlling for baseline
  CIPN-20 sensory subscale (Postma et al 2005). The subscale includes 9 questions, each rated 1-4, and the score ranges from 9-36 with larger values reflecting more severe (worse) symptoms of chemotherapy-induced peripheral neuropathy (CIPN).

OTHER OUTCOMES:
Musculoskeletal function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Leg strength via isokinetic dynamometer test
Cardiovascular function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Distance walked in six-minute walk test
Neuropsychological function | Time point 2 (approx. 6 weeks), controlling for baseline
  Brain connectivity via functional magnetic resonance imaging
Immunological function | Time point 2 (approx. 6 weeks) or time point 3 (approx. 12 weeks), controlling for baseline
  Inflammatory cytokine concentration via ELISA (IL-6, IL-10, etc.)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Maryland, Baltimore, Maryland
  - University of Rochester Medical Center, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Interested researchers may contact the study PI with requests for collaboration.

REFERENCES:
- [Background] Postma TJ, Aaronson NK, Heimans JJ, Muller MJ, Hildebrand JG, Delattre JY, Hoang-Xuan K, Lanteri-Minet M, Grant R, Huddart R, Moynihan C, Maher J, Lucey R; EORTC Quality of Life Group. The development of an EORTC quality of life questionnaire to assess chemotherapy-induced peripheral neuropathy: the QLQ-CIPN20. Eur J Cancer. 2005 May;41(8):1135-9. doi: 10.1016/j.ejca.2005.02.012. Epub 2005 Apr 14. PMID 15911236